CLINICAL TRIAL: NCT01943097
Title: The Evaluation of the 6-[18F]Fluoro-levo-dopa and 123I-MIBG Uptake in the Patients With Neuroblastoma
Brief Title: Evaluation of 18F-dopa and 123I-MIBG Uptake in the Patients With Neuroblastoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200703053M
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Neuroblastic tumors are childhood neoplasms that possess amino acid decarboxylase (AADC) activity and Meta-iodobenzylguanidine(MIBG), they can theoretically be imaged by (18)F-fluorodihydroxyphenylalanine ((18)F-FDOPA) and (123)I-Meta-iodobenzylguanidine((123)I-MIBG) PET, they are new and specific diagnostic and follow-up tools for neuroendocrine tumors. In this study, we explored the accuracy and clinical role of (18)F-FDOPA and (123)I-MIBG PET in neuroblastic tumors.

METHODS:

Patients with tissue-proven neuroblastic tumors receiving (18)F-FDOPA PET or (123)I-MIBG at initial diagnosis or during follow-ups were enrolled. The sensitivity and specificity of (18)F-FDOPA or (123)I-MIBG PET were compared to each other and compared to(18)F-FDG PET, using tumor histology as the standard.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosed by clinical criteria(one of below)

  1. Proved as Neuroblastoma by a pathological section
  2. Bone meta with 24 hrs urine VMA(Vanillylmandelic acid )or HVA (Homovanillic acid) elevated
  3. CT or MRI found tumor around adrenal gland or Neuroblastic tumor
* (2) Age between 0-30 years old，Body weight over 2.5kg
* (3) Signed Inform Consent Form

Exclusion Criteria:

* (1)AST and ALT > 200U/L、Cre > 2.5mg/dl
* (2)Allerg to 18F-dopa、123I-MIBG
* (3)Subject not fit this study(assessed by PI)
* (4)No more need to arrenge PET because disease progress, assessed by VS

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With Neuroblastoma
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2007-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The maximum standardized uptake value and tumor-to-liver uptake ratio | Outcome will be measured in one week after performed.
  The maximum standardized uptake value and tumor-to-liver uptake ratio will be evaluated by specific Nuclear Medicine doctor.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Children Hospital, Taipei, Taiwan, Taiwan